CLINICAL TRIAL: NCT00162201
Title: An Exploratory Study of Changes in Synovial Immune Responses Following BMS-188667 Therapy in Subjects With Active Rheumatoid Arthritis on Background DMARDs Who Have Failed Anti-TNF Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM101-015
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2011-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Parenteral, IV, 500 mg if < 60 kg; 750 mg if > 60 & < 100 kg; 1000 mg if > 100 kg, Monthly, 4 months.
  Other Names: Orencia

SUMMARY:
Study to assess changes in synovial tissue before and after treatment with Abatacept in subjects with RA who remained on their background disease modifying anti-arthritis medications but who have failed previous therapy with anti-TNF (tumor necrosing factor)blocking agents.

ELIGIBILITY:
Inclusion Criteria:

* RA for at least 1 year
* Clear clinical signs of active RA in 1 knee joint
* Meet ARA (1987) criteria for diagnosis of RA and ACR (1991) criteria for RA functional classes I, II, or III
* Inadequate clinical response to a minimum of 3 months of therapy with anti-TNF-blocking agents
* Taking background DMARDs for a minimum of 3 months and at stable doses for at least 28 days

Exclusion Criteria:

* Serious bacterial infection in last 3 months
* History of TB
* History of cancer within 5 years
* Evidence of latent or active bacterial or viral infection
* Intra-articular corticosteroids within 3 months
* Exposure to live vaccines
* Exposure to CTLA4Ig or BMS-188667
* Treatment with immunoadsorption column(s), mycophenolate mofetil, leflunomide, anakinra, cyclosporine, etanercept, adalimumab, infliximab, azathioprine, oral or parenteral gold, D-penacillamine, calcineurin inhibitors, cyclophosphamide or other alkylating agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-10; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Comparison of each subject's synovial tissue markers | at baseline and after 4 months of treatment with abatacept

SECONDARY OUTCOMES:
assess baseline & post treatment synovitis by dynamic gadolinium enhanced MRI; determine concentrations of abatacept in synovial fluid & serum | after 4 months of treatment
assess safety & tolerability of abatacept | administered for 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Leeds, Essex, United Kingdom

REFERENCES:
- [Background] Buch MH, Boyle DL, Rosengren S, Saleem B, Reece RJ, Rhodes LA, Radjenovic A, English A, Tang H, Vratsanos G, O'Connor P, Firestein GS, Emery P. Mode of action of abatacept in rheumatoid arthritis patients having failed tumour necrosis factor blockade: a histological, gene expression and dynamic magnetic resonance imaging pilot study. Ann Rheum Dis. 2009 Jul;68(7):1220-7. doi: 10.1136/ard.2008.091876. Epub 2008 Sep 4. PMID 18772191
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx